CLINICAL TRIAL: NCT07225426
Title: Log2LoseAI: Reinforcement Learning to Create a Framework for Personalizing Financial Incentives
Brief Title: Personalizing Financial Incentives
Acronym: Log2LoseAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Corrine Voils, Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00188990; R34HL170205 (NIH)
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Obesity & Overweight
Keywords: behavioral intervention; obesity; financial incentives; reinforcement learning; artificial intelligence
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized incentives (Experimental): Participants may receive financial incentives for weight loss if their performance suggests they respond to financial incentives.
  Interventions: Behavioral: personalized financial incentives

INTERVENTIONS:
Behavioral: personalized financial incentives — Every week, a reinforcement learning algorithm will process data on weight loss, calorie logging, and incentives earned to predict that their weight loss is positively influenced by incentives.

SUMMARY:
The purpose of this study is to determine the feasibility of providing personalized incentives for dietary self-monitoring and/or interim weight loss to people enrolled in a weight-loss program

DETAILED DESCRIPTION:
In this study, community outpatients will participate in a clinician-facilitated, group-based behavioral weight-loss program for 24 weeks. Dietary self-monitoring data (input by patients via a mobile phone dietary application) and weight data (input by patients via cellular scale) will be collected by a software platform. A reinforcement learning algorithm will use data collected during the trial to predict which participants will respond to a financial incentive. Incentives will be provided to participants predicted to respond, and they will be notified of incentives via text messaging.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to attend virtual baseline and follow-up data collection visits
2. At least 18 years of age
3. Verified obesity as defined as a BMI ≥30 kg/m2
4. Agree to attend 13 biweekly group classes (virtual) delivered by a registered dietitian
5. Agree to review study materials between classes
6. Regular access to an unshared smart phone
7. Reliable access to internet
8. Able to speak and read English
9. Desire to lose weight
10. Able to connect to a video conference call using a smartphone, tablet or computer with a webcam and microphone
11. Ability to download and use Fitbit app daily
12. Have or be willing to create a Gmail address
13. Physical ability to stand on a scale without support

Exclusion Criteria:

1. Weight loss of at least 10lbs in the month prior to screening
2. Weight > 380lbs
3. Currently enrolled or enrolled in the previous month in a clinical, research, or community program focusing on lifestyle change that could affect weight
4. New user of weight loss medication
5. Pregnant, lactating or planning on becoming pregnant during the study
6. History of bariatric procedure or planning to have bariatric procedure in the study timeframe
7. Residing in a nursing home, skilled nursing facility or assisted living facility
8. Impaired hearing
9. Significant dementia, drug or alcohol abuse, or unstable psychiatric illness (e.g., schizophrenia, psychosis)
10. Current treatment for cancer or being treated for cancer (besides basal cell carcinoma or squamous cell) in the last 6 months
11. Use of insulin, sulfonylureas, or meglitinides due to increased risk for hypoglycemia
12. Diuretic medication doses higher than hydrochlorothiazide or chlorthalidone 25 mg daily, furosemide 40 mg daily, torsemide 20 mg daily, bumetanide 1 mg daily, or any use of metolazone; use of potassium-sparing diuretics is acceptable
13. Unstable heart disease in the 6 months prior to screening
14. Chronic kidney disease at stage 4 or higher
15. Exertional chest pain
16. Pain, fainting, or other conditions that prohibit mild/moderate exercise
17. History of ascites requiring paracentesis
18. Inducing vomiting to prevent weight gain or counteract the effects of eating an average of 1 time per week or more in the past 3 months*
19. Not suitable for study participation due to other reasons at the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Screening-to-enrollment ratio | Week 0
  number of potential participants screened for the study/ number of participants who provide a baseline weight for the intervention
Retention for outcomes | 25 weeks
  number of participants who provide a weight at 25 weeks/number of participants who provide a baseline weight for the intervention

SECONDARY OUTCOMES:
Adherence to calorie logging | 24 weeks
  Proportion of weeks participants achieve adequate calorie logging (5 days per week)
Adherence to self-weighing | 24 weeks
  Proportion of weeks participants weigh at least twice per week on a study-provided cellular scale
Body weight | baseline to 25 weeks
  Changes in body weight from baseline to week 25, measured by study-provided cellular scales

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will collect weight data from the cellular-connect scales, calorie logging data from the dietary tracking app, and self-reported survey data including demographics and behavioral measures. Additional data will include binary indicators for whether participants earned an incentive each week of the study and how much they earned, generated by algorithms created by the research team using scale and dietary tracking app data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Scientific data will be available by the earlier of these two time points, as required by the NIH: 1) the date on which the article is first made available in print or electronic format, or 2) the funding period (to include a possible no-cost extension).